CLINICAL TRIAL: NCT00568503
Title: A Partially Blinded, Single-dose, Cross-over Proof of Concept Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of QAX028 Compared to Open-label Tiotropium Bromide (Positive Control) and Placebo in Mild-to-moderate COPD Patients
Brief Title: Safety, Tolerability and Pharmacodynamics of QAX028 Compared to Open-label Tiotropium Bromide and Placebo in Mild-to-moderate Chronic Obstructive Pulmonary Disease (COPD) Patients.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX028A2102
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: COPD
Keywords: COPD/TIOTROPIUM/QAX028
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): QAX028 high dose
  Interventions: Drug: QAX028
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 3 (Active Comparator): Tiotropium bromide
  Interventions: Drug: Tiotropium bromide
- 4 (Active Comparator): QAX028 medium dose
  Interventions: Drug: QAX028
- 5 (Active Comparator): QAX028 low dose
  Interventions: Drug: QAX028

INTERVENTIONS:
Drug: QAX028
  Arms: 1
Drug: Placebo
  Arms: 2
Drug: Tiotropium bromide
  Arms: 3
Drug: QAX028
  Arms: 4
Drug: QAX028
  Arms: 5

SUMMARY:
This will be a single dose Proof-of-Concept study in mild-to-moderate COPD patients. The study will investigate the safety and tolerability of QAX028 as well as the bronchodilatory effects of QAX028 compared to tiotropium and placebo in mild-to-moderate COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 40-75 years with diagnosis of mild or moderate COPD
* Current or X-smokers with a smoking history of >10 pack-years.
* Screening ipratropium post-bronchodilation FEV1 at 1 h post-dose will be greater than 50% of the normal predicted FEV1 value.

Exclusion Criteria:

* Patients who can not comply with the following washout periods for standard

COPD treatments as follows should be excluded:

* Short-acting bronchodilators
* Long-acting bronchodilators
* Inhaled steroids

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and pharmacodynamics of a single dose of QAX028 compared to tiotropium bromide 18μg and to placebo. | throughout the study

SECONDARY OUTCOMES:
The forced expiratory volume in 1 second (FEV1)and time profile using a kinetic pharmacodynamic (KPD) model on single doses of QAX028. Pharmacokinetics of inhaled doses of QAX028. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigative site
Locations (1):
- Novartis Investigator Site, Birkeroed, Denmark